CLINICAL TRIAL: NCT03420794
Title: Optimization of Pre-operative Oral Analgesics in Patients Undergoing Ambulatory Minimally Invasive Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Pamela Frazzini Padilla, Investigator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLA17-099
Record Dates: First submitted 2018-01-24; First posted 2018-02-05 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Hysterectomy; Laparoscopy; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients undergoing total laparoscopic hysterectomy for benign disease who will receive celecoxib 200mg, acetaminophen 1000mg, and gabapentin 600mg by mouth once just prior to surgery.
  Interventions: Other: Timing of pre-operative oral non-narcotic analgesics in relation to minimally invasive hysterectomy
- Study Group (Experimental): Patients undergoing total laparoscopic hysterectomy for benign disease who will receive celecoxib 200mg, acetaminophen 1000mg, and gabapentin 600mg by mouth once 3-4 hours prior to surgery.
  Interventions: Other: Timing of pre-operative oral non-narcotic analgesics in relation to minimally invasive hysterectomy

INTERVENTIONS:
Other: Timing of pre-operative oral non-narcotic analgesics in relation to minimally invasive hysterectomy — Patients will be screened, enrolled, consented, and randomized during the preoperative office encounter, typically occurring within the 30 days prior to surgery. Patients randomized to pre-admission administration (study group) will be provided with a prescription for a one-time dosing of routine oral non-narcotic analgesic medications to be filled at the Cleveland Clinic outpatient pharmacy. Both the study and the control groups will receive written pre-operative instructions. Those patients randomized to the standard practice of administration in the pre-anesthesia unit (control group) will be administered the same medications in the same doses by the nursing staff. Patients in both groups will undergo general anesthesia, orogastric tube placement, and minimally invasive hysterectomy (MIH). Postoperatively, these patients will be observed for differences in PACU narcotic uptake, pain scores, patient satisfaction, and surgical recovery.

SUMMARY:
This is a randomized controlled trial comparing pre-admission administration of routine oral preoperative non-narcotic analgesics with the administration of these medications in the pre-anesthesia care unit per our standard practice. Patients will be screened, enrolled, consented, and randomized during the preoperative office encounter, typically occurring within the 30 days prior to surgery. Patients randomized to pre-admission administration (study group) will be provided with a prescription for a one-time dosing of routine oral non-narcotic analgesic medications to be filled at the Cleveland Clinic outpatient pharmacy. Both the study and the control groups will receive written pre-operative instructions. Those patients randomized to the standard practice of administration in the pre-anesthesia unit (control group) will be administered the same medications in the same doses by the nursing staff.

Patients in both groups will undergo general anesthesia, orogastric tube placement, and minimally invasive hysterectomy (MIH). Post-operatively, patient pain will be assessed via NRS at standard intervals and treated with narcotics. Amount of total intravenous (IV) and oral (PO) narcotics given during PACU stay will be documented in the medication administration record (MAR) within the electronic medical record (EMR) and later converted into oral morphine equivalents (OME). Pain will be assessed via NRS on discharge and documented.

Patients will be emailed on POD10 a survey to rate their satisfaction with their medication administration regimen on a 5-point Likert scale. Participants will also be asked to complete a thirteen-point surgical recovery scale (SRS) to evaluate their functional recovery from MIH.

Patient participation will conclude after completion of the patient satisfaction survey and SRS. A maximum of 58 patients will be enrolled into the study, as we aim to randomize 26 patients to each arm.

DETAILED DESCRIPTION:
This is a randomized controlled trial comparing pre-admission administration of routine oral preoperative non-narcotic analgesics with the administration of these medications in the pre-anesthesia care unit per our standard practice. Patients will be screened, enrolled, consented, and randomized during the preoperative office encounter, typically occurring within the 30 days prior to surgery. Patients randomized to pre-admission administration (study group) will be provided with a prescription for a one-time dosing of routine oral non-narcotic analgesic medications to be filled at the Cleveland Clinic outpatient pharmacy. Both the study and the control groups will receive written pre-operative instructions. Those patients randomized to the standard practice of administration in the pre-anesthesia unit (control group) will be administered the same medications in the same doses by the nursing staff.

Patients in both groups will undergo general anesthesia, orogastric tube placement, and minimally invasive hysterectomy (MIH). Post-operatively, patient pain will be assessed via NRS at standard intervals and treated with narcotics. Amount of total intravenous (IV) and oral (PO) narcotics given during PACU stay will be documented in the medication administration record (MAR) within the electronic medical record (EMR) and later converted into oral morphine equivalents (OME). Pain will be assessed via NRS on discharge and documented.

Patients will be emailed on POD10 a survey to rate their satisfaction with their medication administration regimen on a 5-point Likert scale. Participants will also be asked to complete a thirteen-point surgical recovery scale (SRS) to evaluate their functional recovery from MIH.

Patient participation will conclude after completion of the patient satisfaction survey and SRS. A maximum of 58 patients will be enrolled into the study, as we aim to randomize 26 patients to each arm.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be women, at least 18 years of age
2. Subjects must be undergoing minimally invasive hysterectomy for benign indications
3. Subjects must be capable of giving informed consent
4. Subjects must be English-language speaking. This is required as the validated surgical recovery surveys utilized in this protocol have not been validated in any language other than English.

Exclusion Criteria:

1. Subjects may not have a history of chronic pain
2. Subjects may not have a history of chronic use of pain medication
3. Subjects may not have an allergy or medical contraindication to the preoperative non-narcotic analgesics or to opioid pain medication
4. Subjects must not have been previously diagnosed with gastroparesis, impaired gastric emptying, personal history of gastric bypass, or any neuromuscular degenerative disease. Subjects previously diagnosed with gastro-esophageal reflux are permitted.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 58 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Immediate post-operative opioid requirement | On the date of surgery from the time surgery was completed to the time the patient is discharged from the post-anesthesia care unit, up to 24 hours
  To determine the immediate post-operative opioid requirement

SECONDARY OUTCOMES:
Patient Satisfaction | 10-14 days after surgery
  To evaluate patient satisfaction via online survey with each preemptive multimodal analgesic regimen. Patient satisfaction will be evaluated via online survey with each pain regimen using a 5 point Likert scale (5 being extremely satisfied and 1 being extremely dissatisfied). The mean score in each group will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No